CLINICAL TRIAL: NCT06382207
Title: Effectiveness of the Eko Digital Stethoscope in Capturing Infant Electrocardiograms
Brief Title: Effectiveness of the Eko Digital Stethoscope in Capturing Infant ECGs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HM20029298
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Tachyarrhythmia
Keywords: Infant Tachyarrhythmia; Cardiac Rhythm; Digital Stethoscope
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Intervention Model Description: This proof-of-concept study will enroll infants, defined as individuals <1 year of age. It will assess the feasibility and effectiveness of a physician and parent/caregiver in using the Eko DUO and CORE 500 to capture ECGs in patients <10 kg in a clinic and home setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital Stethoscopes to measure neonatal tachyarrhythmias (Other): Parental caregivers of infant research subjects are trained to use technology (digital stethoscopes) to decrease stress and unnecessary trips to the emergency room.
  Interventions: Device: Eko Duo electronic stethoscope; Device: CORE 500 electronic stethoscope

INTERVENTIONS:
Device: Eko Duo electronic stethoscope — A digital stethoscope with 1-lead electrocardiogram (ECG), the DUO, which pairs with a mobile application that allows the clinician to further engage with the device during and after a clinical visit. The application enables the clinician to visualize the sounds and electrical signals coming from the device in real time.
Device: CORE 500 electronic stethoscope — The CORE 500 has 3 electrodes that produce a 3 lead ECG, which can be viewed through the Eko app. The CORE 500 also has a user interface screen which provides a number of functions including confirming when all three electrodes have good skin contact, showing a single lead ECG wave, providing heart rate, allowing the user to switch between audio modes, allowing the user to take recordings, and providing AI analysis results for recordings.

SUMMARY:
When a newborn is diagnosed with tachyarrhythmia, they are generally started on medical therapies, most commonly a beta-blocker, while being observed in an inpatient setting. In most academic institutions, current practice is to provide parental teaching on use of a stethoscope to auscultate their child when there is suspicion for distress, in addition to requiring cardiopulmonary resuscitation (CPR) classes. Fortunately, newer technologies have emerged that allow for capture of cardiac rhythm that may provide a buffer between the infant and the emergency room.

DETAILED DESCRIPTION:
Tachyarrhythmias which would prompt an emergent call to the pediatric cardiologist following the child, along with simultaneous transportation towards the nearest, preferably pediatric, emergency room. In reality, parental caregivers may be blinded by their personal anxiety in caring for their child with a tachyarrhythmia, and their interpretation or ability to count their child's heart beats may not be accurate. This in turn, can result in unnecessary calls and visits to the emergency room which increase their utilization in addition to piling onto the already astounding cost of healthcare in the United States. Fortunately, newer technologies have emerged that allow for capture of cardiac rhythm that may provide a buffer between the infant and the emergency room. Eko manufactures a digital stethoscope with 1-lead electrocardiogram (ECG), the DUO, which pairs with a mobile application that allows the clinician to further engage with the device during and after a clinical visit. The application enables the clinician to visualize the sounds and electrical signals coming from the device in real time.

Currently, the DUO is cleared for use on patients greater than or equal to 10 kg. This device may have additional clinical utility in pediatric patients <10 kg when used by either a physician or a parent/caregiver at home for remote patient monitoring. The CORE 500 may also have clinical utility in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age <1 year
* No previous diagnosis of arrhythmia
* Parent/caregiver can provide informed consent
* Parent/caregiver can speak and understand simple English

Exclusion Criteria:

* Age ≥ 1 year
* Patient has a pacemaker or implantable cardioverter defibrillator (ICD)
* Parent/caregiver is unwilling or unable to provide informed consent
* Parent/caregiver is unable to speak and understand English

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of good-quality ECG recordings taken by physicians, for DUO and for CORE 500 | Baseline Visit
  Number and proportion of good-quality ECG recordings taken by physicians, for DUO and for CORE 500. A "good-quality" ECG recording is defined as one where the tracing is clear enough and with sufficient amplitude to define the p-wave, QRS complex, and t-wave, beyond a reasonable doubt, to allow determination of the patient's cardiac rhythm, by two independent pediatric electrophysiologists and a pediatric cardiologist.
Number and proportion of good-quality ECG recordings taken by parents/caregivers, with a physician present in the exam room using the CORE 500 | Baseline Visit
  Number and proportion of good-quality ECG recordings taken by parents/caregivers, with a physician present in the exam room, for CORE 500. A "good-quality" ECG recording is defined as one where the tracing is clear enough and with sufficient amplitude to define the p-wave, QRS complex, and t-wave, beyond a reasonable doubt, to allow determination of the patient's cardiac rhythm, by two independent pediatric electrophysiologists and a pediatric cardiologist.
Number and proportion of good-quality ECG recordings taken by parents/caregivers, with a physician absent from the exam room, for CORE 500 | Baseline Visit
  Number and proportion of good-quality ECG recordings taken by parents/caregivers, with a physician absent from the exam room, for CORE 500. A "good-quality" ECG recording is defined as one where the tracing is clear enough and with sufficient amplitude to define the p-wave, QRS complex, and t-wave, beyond a reasonable doubt, to allow determination of the patient's cardiac rhythm, by two independent pediatric electrophysiologists and a pediatric cardiologist.
Number and proportion of good-quality ECG recordings taken by parents/caregivers, at home, for CORE 500 only | At end of study (two weeks)
  Number and proportion of good-quality ECG recordings taken by parents/caregivers, at home, for CORE 500. A "good-quality" ECG recording is defined as one where the tracing is clear enough and with sufficient amplitude to define the p-wave, QRS complex, and t-wave, beyond a reasonable doubt, to allow determination of the patient's cardiac rhythm, by two independent pediatric electrophysiologists and a pediatric cardiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Snyder, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States